CLINICAL TRIAL: NCT02202044
Title: Adjuvant Sequential Intravesical BCG (Bacillus Calmette-Guérin) and Electromotive Mitomycin-C (EMDA/MMC) After Transuretheral Resection (TUR) in Patients With Primary High Risk Non-Muscle Invasive Transitional Cell Carcinoma of the Bladder
Brief Title: Sequential Intravesical Bacillus Calmette-Guérin and Electromotive Mitomycin-C After Transuretheral Resection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The institution was requiring extensive changes to the protocol
Sponsor: University of Colorado, Denver (Other)
Collaborators: Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-1359.cc
Record Dates: First submitted 2014-07-24; First posted 2014-07-28 (Estimated); Results first posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-05

CONDITIONS: Bladder Carcinoma
Keywords: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intravesical BCG and EMDA/MMC (Experimental): Patients are assigned one course of treatment per week for 6 weeks of Intravesical Intravesical BCG and EMDA/MMC
  Interventions: Device: Intravesical BCG and EMDA/MMC

INTERVENTIONS:
Device: Intravesical BCG and EMDA/MMC — Patients are assigned one course of treatment per week for 6 weeks with sequential 'Intravesical instillation of sequential Bacillus Calmette-Guérin (BCG) and Electromotive Drug Administration /Mitomycin-C

SUMMARY:
The primary objective of the study is to assess the bladder cancer recurrence free rate, according to a phase II pilot study, of intravesical instillation of sequential BCG and EMDA/MMC after TUR. The study is designed as a one-sample investigation: the outcome measure is disease recurrence rate. Follow up will continue up to 5 years.

For sample size determination, disease recurrence rate will be compared with literature data of recurrence rate obtained in standard BCG alone administration (Lamm's protocol).

DETAILED DESCRIPTION:
TURBT (TransUrethral Resection of Bladder Tumor)

Prior to enrolment, all patients must sign a consent form and will have a Complete Blood Count (CBC), Basic Metabolic Panel (BMP) and a Urinalysis (UA) performed. The patients White Blood Count (WBC) must be greater than 4.0 10^9/L and platelet count greater than 150 10^9/L to receive drug.

Week 1, 2, 4, 5, 7 and 8: BCG instillation: 50 mg wet weight (10•2±9•0x108 colony-forming units) BCG Connaught substrain. Lyophilised (ie, freeze-dried) BCG are suspended in 50 ml bacteriostatic-free 0.9% Sodium Chloride (NaCl) solution. After bladder draining, the suspension is infused intravesically through a 14 Fr Foley catheter and retained in the bladder for 60-90 min; bladder emptying is followed by catheter removal.

Week 3, 6 and 9: A Foley catheter is inserted and the bladder is carefully drained. 40 mg MMC dissolved in 100 ml NaCl 0.9% solution are instilled intravesically through the electrode catheter by gravity and retained in the bladder for 30 min, while 23 mA for 30 min pulsed electric current is given externally. Two dispersive cathode electrodes are placed on lower abdominal skin after degreasing with alcohol. The bladder is then emptied and the catheter removed. Patients are assigned one course of treatment per week for 6 weeks with sequential BCG and EMDA/MMC. Two BCG instillations and one EMDA/MMC instillation constitute one cycle for a total of two cycles.

A CBC and basic metabolic panel (BMP) will be performed weekly and at the beginning of each cycle. Prior to dosing with mitomycin C at week 3, a CBC will be performed and also at weeks 4 and 5 if the CBC has changed. A UA will be performed prior to each intravesicular instillation.

Maintenance treatment of eMMC will be given at month 3, 4, 6, 7, 9 and 10 (after last dose of BCG of the initial treatment). Maintenance of BCG will be given around month 5, 8, and 11. CBC, BMP, UA, and a history/physical (H&P) will be performed before each EMDA/MMC procedure. UA and a H&P will be performed before each BCG.

ELIGIBILITY:
Inclusion Criteria:

* After a restaging TURBT patients with histologically proven primary high grade (grade3) and/or pT1 transitional cell carcinoma of the bladder, with or without pTis and pTis alone are regarded as being at high risk for tumour recurrence and progression.
* Patients may enroll in this study if they are thought to have no residual disease after TURBT.
* Age 18 years or over
* Adequate bone-marrow reserve- ECOG performance status between 0 and 2
* Patients who are known PPD positive will be screened for active tuberculosis prior to starting treatment with BCG.

Exclusion Criteria:

* known allergy to BCG or MMC
* prior systemic infection with BCG
* prior or concomitant urothelial tumours of the upper urinary tract or urethra
* previous muscle-invasive (ie, stage T2 or higher) transitional-cell carcinoma of the bladder
* bladder capacity of less than 200 ml
* untreated urinary-tract infection
* severe systemic infection (ie, sepsis)
* known HIV-positivity; therapy with immunosuppressive agents
* urethral strictures that would prevent endoscopic procedures and repeated catheterisation
* upper urinary tract disease (eg, vesicoureteral reflux or urinary-tract stones) that would make multiple transurethral procedures a risk
* previous radiotherapy to the pelvis
* other concurrent chemotherapy
* treatment with radiotherapy-response or biological-response modifiers
* history of tuberculosis;
* other malignant diseases within 5 years of trial registration (except for adequately treated basal-cell or squamous cell skin cancer, in situ cervical cancer and any other cancer from which patients has been disease-free for 3 years);
* pregnancy or nursing
* psychological, familial, sociological, or geographical factors that would preclude study participation.
* Patients with implantable or wearable electrical devices will be excluded from this study.
* Patients with active tuberculosis

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-02-24 (Actual); Primary Completion 2016-05-11 (Actual); Study Completion 2016-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shandra Wilson, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - Donald Lam, MD, Phoenix, Arizona
  - University of Colorado Denver, Aurora, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated before participants finished treatment and the PI is no longer in the institution to provide information for results reporting. No results information is available.
Period: Overall Study
Arm/Group | Intravesical BCG and EMDA/MMC
Started | 0
Completed | 0
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated before participants finished treatment and the PI is no longer in the institution to provide information for results reporting. No results information is available
Arm/Group | Intravesical BCG and EMDA/MMC
Number analyzed (Participants) | 0
Age, Continuous
Sex: Female, Male
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: To Assess Disease Recurrence Rate
Time Frame: 5 years
Population: as for baseline characteristics
Arm/Group | Intravesical BCG and EMDA/MMC
Number analyzed (Participants) | 0

2. Secondary Outcome: To Compare Complete Response Rates at 3 and 6 Months in Patients With Carcinoma in Situ.
Time Frame: 5 years
Population: as for baseline characteristics
Arm/Group | Intravesical BCG and EMDA/MMC
Number analyzed (Participants) | 0

3. Other Pre Specified Outcome: To Compare the Qualitative and Quantitative Toxicities of Experimental Regimens in These Patients.
Time Frame: 5 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: To Assess Long-term Morbidity in the Study Group, as Defined by Requirement for Fewer TURBTs, Courses of Traditional Intravesical Therapies, and Surveillance Cystoscopies Over 5 Years (Cost-effectiveness)
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: The study was terminated before participants finished treatment and the PI is no longer in the institution to provide information for results reporting. No results information is available.
Description: The study was terminated before participants finished treatment and the PI is no longer in the institution to provide information for results reporting. No results information is available.
Arm/Group | Intravesical BCG and EMDA/MMC
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes